CLINICAL TRIAL: NCT04766177
Title: Role of Bumetanide in Treatment of Autism Spectrum Disorder in Children
Brief Title: Role of Bumetanide in Treatment of Autism
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: autism
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Bumetanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bumetanide group (Experimental): Bumetanide a dose of 0.5 mg twice per day
  Interventions: Drug: Bumetanide
- Placebo (Placebo Comparator): Placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bumetanide — bumetanide 0.5 mg twice daily
  Other Names: burinex
  Arms: bumetanide group
Drug: Placebo — placebo tablets twice daily
  Other Names: Placebo treatment
  Arms: Placebo

SUMMARY:
Role of bumetanide in Autism

DETAILED DESCRIPTION:
Role of Bumetanide in Treatment of Autism spectrum disorder in children

ELIGIBILITY:
Inclusion Criteria:

1. All patients with ASD diagnosed by CARS rating Scale⩾30.
2. Age of patients range between (3-12) years.

Exclusion Criteria:

* Patients with ASD associated with neurological antecedents (including epilepsies and febrile seizures), hepatic, renal dysfunction or electrocardiogram abnormalities and syndromatic children(Rett).

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with improved CARS score | 6 months
  the patients with improved CARS score

CONTACTS AND LOCATIONS:
Overall Officials: Osama Elagamy, Prof, Principal Investigator — Pediatrics Department- Kafr-Elsheikh University; Abeer Salamah, Dr, Study Director — Pediatrics Department- Kafr-Elsheikh University; Esraa Shaker, Msc, Principal Investigator — Pediatrics Department- Kafr-Elsheikh University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No